CLINICAL TRIAL: NCT06229509
Title: Study of Cytokine Response During Exercise Dyspnea in Patients With Chronic Obstructive Pulmonary Disease (COPD). Effect of Body Composition
Brief Title: Study of the Cytokine Response During Exercise Dyspnea in Patients With Chronic Obstructive Pulmonary Disease (COPD). Effect of Body Composition
Acronym: CYTODINE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: AOI 2022 ROLLAND DEBORD
Record Dates: First submitted 2024-01-09; First posted 2024-01-29 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Chronic Obstructive Pulmonary Disease Severe; Dyspnea
Keywords: Cytokines; Myokines; Adipokines; Exercise; Noninvasive Ventilation; Sarcopenia
MeSH Terms: conditions — Dyspnea; Motor Activity; Sarcopenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Effective noninvasive ventilation (Experimental): Alleviate dyspnea (lower Borg Score by 2 points)
  Interventions: Device: Effective noninvasive ventilation
- Sham noninvasive ventilation (Sham Comparator)
  Interventions: Device: Sham noninvasive ventilation

INTERVENTIONS:
Device: Effective noninvasive ventilation — Noninvasive ventilation set to alleviate dyspnea Inspiratory aid set according to a preliminary test (aiming for a diminution of 2 points in Borg score)
  Arms: Effective noninvasive ventilation
Device: Sham noninvasive ventilation — Noninvasive ventilation set with an insufficient inspiratory aid to alleviate dyspnea
  Arms: Sham noninvasive ventilation

SUMMARY:
Dyspnea, more commonly known as breathlessness, is a symptom found in the majority of patients with chronic obstructive pulmonary disease (COPD), with a major impact on quality of life and mortality.

COPD is a chronic inflammatory disease of the bronchi, affecting 8% of the French population (more than 3 million people). By 2030, it will be the third leading cause of death worldwide. Effective management of dyspnea in these patients is a priority.

In patients with severe COPD, physical exertion increases the workload of breathing, leading to dyspnea. At the same time, the respiratory muscles and fatty cells release cytokines, myokines and adipokines - a group of proteins involved in the inflammatory response. In addition, 15% of COPD patients suffer from sarcopenia (loss of muscle mass and strength) which increases respiratory effort and dyspnea.

Our research project aims to study the effect of dyspnea relief in COPD patients on cytokine, myokine and adipokine levels, taking into account the presence of sarcopenia. Indeed, it is possible to alleviate the workload of the respiratory muscles during exercise by means of respiratory assistance.

The ultimate goal is a better understanding of dyspnea mechanisms, to enable the development of cytokine-targeted therapies and improve quality of life and survival in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patient affiliated to a social security scheme.
* Patient capable of giving free, informed, written and signed consent.
* Male gender
* Severe COPD (Chronic Obstructive Pulmonary Disease) diagnosed according to GOLD criteria, in a stable state, with a forced expiratory volume (FEV1) from 30 to 50% of the predicted value (measured within one year during respiratory function tests (RFT)
* History of smoking >10 pack-years with cessation of smoking for more than 12 months.
* Patient judged by the investigator to be able to tolerate inspiratory pressure during a preliminary cycling exercise test.

Exclusion Criteria:

* Severe anxiety disorders, assessed by the STAY Y-B form questionnaire; a score above 65 indicates very high day-to-day anxiety.
* Patient under guardianship/trusteeship/supervision of justice
* Chronic hypercapnia at rest (CO2 arterial pressure ≥ 50mmHg)
* Chronic use of non-invasive ventilation
* Known pulmonary hypertension
* Chronic administration of oral corticosteroids
* Unstable heart disease

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2024-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Variation in exercise-induced release of cytokines IL-1, IL-6, IL-8, IL-10 and TNF-alpha plasma concentrations (pg/mL) between the two ventilatory conditions (sham and effective) | At rest = baseline / right after the end of exercice / 45 minutes after the end of exercice
Variation in exercise-induced release of adipokines adiponectin and leptin concentrations (pg/mL) between the two ventilatory conditions (sham and effective) | At rest = baseline / right after the end of exercice / 45 minutes after the end of exercice

SECONDARY OUTCOMES:
For each ventilatory condition, study of correlation between dyspnea descriptors (Borg scale score, Multidimensional Dyspnea Profil score) and cytokines, adipokines and myokines plasma concentrations (pg/mL) | At rest = baseline / right after the end of exercice / 45 minutes after the end of exercice
For each ventilatory condition, study of correlation between muscle mass (kg) and cytokines, adipokines and myokines plasma concentrations (pg/mL). | At rest = baseline / right after the end of exercice / 45 minutes after the end of exercice
For each ventilatory condition, study of correlation between fat mass (kg) and cytokines, adipokines and myokines plasma concentrations (pg/mL). | At rest = baseline / right after the end of exercice / 45 minutes after the end of exercice

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

IPD SHARING:
Plan to Share IPD: No